CLINICAL TRIAL: NCT03239197
Title: An Exploratory Study to Evaluate the Transfer of the Maternal Microbial Consortia to Infants During and Following Birth
Brief Title: Project SHARE (motherS Have All the Right microbEs)
Status: Withdrawn | Type: Observational
Why Stopped: Sponsor request
Sponsor: Kimberly-Clark Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: 500-16-0004
Record Dates: First submitted 2017-08-01; First posted 2017-08-03 (Actual); Last update posted 2017-12-12 (Actual); Status verified 2017-12

CONDITIONS: Microbiota

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Biospecimen Retention: None Retained — staphlococci isolates
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- mother infant pair: mother infant pair, singleton infant, vaginal birth

SUMMARY:
This is an exploratory study designed to collect microbial samples from several body locations from 6 pairs of mothers and their newborn infants at various time points.

ELIGIBILITY:
Inclusion Criteria:

* Mother- pregnant female, singleton infant
* Infant- vaginal birth, breastfeeding as primary source of nutrition

Exclusion Criteria:

* Mother- antibiotic, steroid or antimicrobial use
* Infant- antibiotic, steroid or antimicrobial use

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: pregnant mothers and their infants, planning a vaginal birth and breastfeeding as primary source of nutrition
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2017-09-05 (Actual); Primary Completion 2018-03 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Maternal staphylococci is transferred to infant during and following birth. | 6 weeks
  presence of maternal staphylococci strain in infant

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Welter, MD, Principal Investigator — Marshfield Clinic
Locations (1):
- Marshfield Clinic, Marshfield, Wisconsin, United States

REFERENCES:
- [Background] Costello EK, Lauber CL, Hamady M, Fierer N, Gordon JI, Knight R. Bacterial community variation in human body habitats across space and time. Science. 2009 Dec 18;326(5960):1694-7. doi: 10.1126/science.1177486. Epub 2009 Nov 5. PMID 19892944
- [Background] Dowd SE, Sun Y, Wolcott RD, Domingo A, Carroll JA. Bacterial tag-encoded FLX amplicon pyrosequencing (bTEFAP) for microbiome studies: bacterial diversity in the ileum of newly weaned Salmonella-infected pigs. Foodborne Pathog Dis. 2008 Aug;5(4):459-72. doi: 10.1089/fpd.2008.0107. PMID 18713063
- [Background] Capone KA, Dowd SE, Stamatas GN, Nikolovski J. Diversity of the human skin microbiome early in life. J Invest Dermatol. 2011 Oct;131(10):2026-32. doi: 10.1038/jid.2011.168. Epub 2011 Jun 23. PMID 21697884
- [Background] Mueller NT, Bakacs E, Combellick J, Grigoryan Z, Dominguez-Bello MG. The infant microbiome development: mom matters. Trends Mol Med. 2015 Feb;21(2):109-17. doi: 10.1016/j.molmed.2014.12.002. Epub 2014 Dec 11. PMID 25578246
- [Background] Johnson CL, Versalovic J. The human microbiome and its potential importance to pediatrics. Pediatrics. 2012 May;129(5):950-60. doi: 10.1542/peds.2011-2736. Epub 2012 Apr 2. PMID 22473366
- [Background] Madan JC, Farzan SF, Hibberd PL, Karagas MR. Normal neonatal microbiome variation in relation to environmental factors, infection and allergy. Curr Opin Pediatr. 2012 Dec;24(6):753-9. doi: 10.1097/MOP.0b013e32835a1ac8. PMID 23111681